CLINICAL TRIAL: NCT00873548
Title: Treatment of Unstable Trochanteric Fractures With the Proximal Femoral Nail - Antirotation Asia - A Prospective Multicenter Case Series
Brief Title: Treatment of Unstable Trochanteric Fractures With the Proximal Femoral Nail - Antirotation (PFNA)-Asia
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: Synthes Inc. (Industry)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: PFNA_Asia
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2013-01

CONDITIONS: Trochanteric Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PFNA_Asia treated
  Interventions: Device: PFNA-Asia

INTERVENTIONS:
Device: PFNA-Asia — The operation is performed under regional or general anesthesia and involves the following main steps:
  1. Positioning of the patient
  2. Definition of the CCD-angle
  3. Fracture reduction
  4. Determination of the nail diameter
  5. Incision
  6. Insertion of the device

SUMMARY:
The primary objective of this prospective multicenter study is to assess any fracture fixation complication and revision rates during the clinical use of the Proximal Femoral Nail Antirotation Asia (PFNA Asia) for the treatment of unstable trochanteric fractures.

DETAILED DESCRIPTION:
From several studies, e.g. on hip prostheses, it is known that the Asian population has other geometric proportions than Caucasians, e.g. Japanese woman have shorter femoral necks, smaller femoral neck angles and a more anterior bowing of the shaft than white Americans. This was one of the reasons for the development of a new PFNA Asia with adapted sizes and geometry. No controlled clinical data are available whether the rate of mismatch and mismatch-related complications could be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older
* Patients with isolated, unstable, closed trochanteric fractures, classified as AO 31-A2 or AO 31-A3
* Definitive primary fracture treatment with PFNA Asia within 7 days sustaining the fracture (conversion from an external fixator to the PFNA Asia as an emergency procedure within the first week after the accident is allowed)
* Signed written informed consent (by the subjects or legal guardian) and agreement to attend the planned follow-ups
* Willing and able to comply with the post-operative management program
* Able to understand and read country national language at an elementary level

Exclusion Criteria:

* Pathologic fracture
* Patients or legal guardian refusing to sign the informed consent form
* Patients with previous implants on the fractured hip and femur
* Drug or alcohol abuse
* Active malignancy
* ASA class V and VI
* Patients who are bed-ridden or wheel-chair ridden prior to injury event
* Neurological disorders and psychiatric disorders that would preclude reliable assessment (e.g., Parkinson disease, Multiple sclerosis, severe depression)
* Patients who have participated in any other device or drug related clinical trial within the previous month

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with acute trochanteric fractures at surgery/ orthopedic departments
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2007-11; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Bone/fracture- or implant/surgery-related fracture fixation complication events | 6 and 12 weeks, 6 and 12 months

SECONDARY OUTCOMES:
Mismatch | Perioperatively
Soft tissue/wound -related or general complications | 6 and 12 weeks, 6 and 12 months
Health-related quality of life assessed by the generic SF-36-instrument and EQ-5D | Baseline, 6 and 12 months
Walking ability (Parker mobility score) | Baseline, 6 and 12 months
Range of motion (ROM) | 6 and 12 weeks, 6 and 12 months
Mortality | 6 and 12 weeks, 6 and 12 months
Surgery details and postoperative treatment | till 12 weeks after surgery
Length of hospital stay | till 12 weeks after surgery
Capacity to return to pre-residential status | 12 weeks
Bone consolidation and anatomical restoration | 6 and 12 weeks, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Sawaguchi, MD, Principal Investigator — Toyama Municipal Hospital
Locations (1):
- Toyama Municipal Hospital, Toyama, Japan

REFERENCES:
- [Background] Schipper IB, Marti RK, van der Werken C. Unstable trochanteric femoral fractures: extramedullary or intramedullary fixation. Review of literature. Injury. 2004 Feb;35(2):142-51. doi: 10.1016/s0020-1383(03)00287-0. PMID 14736471
- [Background] Nakamura T, Turner CH, Yoshikawa T, Slemenda CW, Peacock M, Burr DB, Mizuno Y, Orimo H, Ouchi Y, Johnston CC Jr. Do variations in hip geometry explain differences in hip fracture risk between Japanese and white Americans? J Bone Miner Res. 1994 Jul;9(7):1071-6. doi: 10.1002/jbmr.5650090715. PMID 7942154
- [Background] Simmermacher RK, Ljungqvist J, Bail H, Hockertz T, Vochteloo AJ, Ochs U, Werken Cv; AO - PFNA studygroup. The new proximal femoral nail antirotation (PFNA) in daily practice: results of a multicentre clinical study. Injury. 2008 Aug;39(8):932-9. doi: 10.1016/j.injury.2008.02.005. Epub 2008 Jun 25. PMID 18582887
- [Background] Simmermacher RK, Bosch AM, Van der Werken C. The AO/ASIF-proximal femoral nail (PFN): a new device for the treatment of unstable proximal femoral fractures. Injury. 1999 Jun;30(5):327-32. doi: 10.1016/s0020-1383(99)00091-1. PMID 10505125